CLINICAL TRIAL: NCT07081542
Title: Comparative Analysis of Hearing Outcomes: Robotic vs. Manual Insertion of Cochlear Implants
Status: Not yet recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: AdventHealth (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: 2269273
Record Dates: First submitted 2025-05-30; First posted 2025-07-23 (Actual); Last update posted 2026-01-02 (Actual); Status verified 2025-05

CONDITIONS: Sensorineural Hearing Loss; Bilateral Hearing Loss; Cochlear Implantation; Hearing Disorders; Hearing Disorders and Deafness; Inner Ear Disorders; Hearing Impairment
Keywords: Cochlear Implant; Robotic Cochlear Implant Insertion; Hearing Performance; Speech Perception; Electrocochleography; Hearing Rehabilitation; Postoperative Hearing Outcomes; Minimally Invasive ENT Surgery
MeSH Terms: conditions — Hearing Loss, Sensorineural; Hearing Loss, Bilateral; Hearing Disorders; Deafness; Vestibular Diseases; Hearing Loss

STUDY DESIGN:
Who Masked: Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: Yes | US Export: No

ARMS (2):
- Robotic-Assisted Cochlear Implant Insertion (Experimental): Surgical technique using robotic assistance (IotaSoft system) to perform the cochlear implant electrode array insertion into the cochlea.
  Interventions: Device: IotaSoft Robotic Insertion System
- Manual Cochlear Implant Insertion (Active Comparator): Standard surgical technique for inserting the cochlear implant electrode array without robotic assistance. This represents the standard of care method.
  Interventions: Procedure: Manual Cochlear Implant Insertion

INTERVENTIONS:
Device: IotaSoft Robotic Insertion System — The IotaSoft robotic insertion device is an FDA-approved tool designed to provide precise and controlled insertion of the cochlear implant electrode array to minimize trauma during implantation.
  Arms: Robotic-Assisted Cochlear Implant Insertion
Procedure: Manual Cochlear Implant Insertion — Standard surgical technique for manually inserting the cochlear implant electrode array. This method reflects the current standard of care without the assistance of robotic tools.
  Arms: Manual Cochlear Implant Insertion

SUMMARY:
This research study is evaluating two different methods of cochlear implant (CI) insertion - robotic-assisted insertion and manual insertion - to better understand how they affect hearing outcomes. Participants in this study will be randomly assigned to receive their cochlear implant using one of these two techniques. Both methods are performed in a standard operating room by qualified surgeons, and both are considered safe and approved for use.

The main goal is to compare how well participants hear one year after surgery based on the insertion method used. The study will also look at things like surgical time, inner ear health, and how the hearing nerve responds. All participants will receive the same type of cochlear implant device and follow-up care.

This study may help guide future surgical techniques and improve outcomes for individuals receiving cochlear implants.

ELIGIBILITY:
Inclusion Criteria:

* Cochlear implant candidates >18 years of age
* LFPTA (125Hz, 250Hz, 500Hz) <80dB

Exclusion Criteria:

* Pediatric patients (below the age of 18)
* LFPTA (125Hz, 250Hz, 500Hz) >80dB
* Revision cases
* Severe comorbidities that contraindicate surgery.
* Preexisting cochlear anomalies.
* Do not speak English or Spanish

Ages: 18 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 32 (Estimated)
Dates: Start 2026-01-01 (Estimated); Primary Completion 2027-01-31 (Estimated); Study Completion 2027-01-31 (Estimated)

PRIMARY OUTCOMES:
Change in Low-Frequency Pure Tone Average (LFPTA) | Baseline (pre-op) to 12 months post-activation
  Change in unaided pure tone thresholds at 125, 250, and 500 Hz from baseline to 12 months post-activation. The average of these frequencies will be computed for each participant.
Speech Recognition Using CNC Word Test | 3, 6, and 12 months post-activation
  Participants' ability to recognize individual spoken words will be assessed using the Consonant-Nucleus-Consonant (CNC) word test in both quiet and noise conditions. Outcome is based on the percent of key words correctly repeated.
Speech Recognition Using AzBio Sentence Test | 3, 6, and 12 months post-activation
  Participants' ability to recognize spoken sentences will be assessed using the AzBio sentence test in quiet and noise. Outcome is based on the percent of key words correctly repeated in standardized sentence lists.
Degree of Low-Frequency Hearing Preservation | Baseline to 12 months post-activation
  Subjects will be categorized based on change in LFPTA into:
  * Full preservation (<15 dB loss)
  * Partial preservation (15-30 dB loss)
  * Significant loss (>30 dB loss)

SECONDARY OUTCOMES:
Impedance Measurements | CI activation (6-8 weeks post-op)
  To assess device function and consistency over time by measuring electrical impedance (in kilo-ohms, kΩ) of cochlear implant electrodes following either robotic or manual insertion. Impedance will be recorded at activation. Lower and more stable impedance values are expected to indicate better electrode-tissue interface and improved device function. The hypothesis is that robotic cochlear implantation will result in lower and more consistent impedance values compared to manual insertion.

CONTACTS AND LOCATIONS:
Locations (1):
- AdventHealth Celebration, Kissimmee, Florida, United States

IPD SHARING:
Plan to Share IPD: No
We will not be sharing information from this study.

REFERENCES:
- [Background] Barriat S, Peigneux N, Duran U, Camby S, Lefebvre PP. The Use of a Robot to Insert an Electrode Array of Cochlear Implants in the Cochlea: A Feasibility Study and Preliminary Results. Audiol Neurootol. 2021;26(5):361-367. doi: 10.1159/000513509. Epub 2021 Apr 26. PMID 33902040
- [Background] Gersdorff G, Peigneux N, Duran U, Camby S, Lefebvre PP. Impedance and Functional Outcomes in Robotic-Assisted or Manual Cochlear Implantation: A Comparative Study. Audiol Neurootol. 2025;30(1):80-88. doi: 10.1159/000540577. Epub 2024 Aug 23. PMID 39182488
- [Background] Heuninck E, Van de Heyning P, Van Rompaey V, Mertens G, Topsakal V. Audiological outcomes of robot-assisted cochlear implant surgery. Eur Arch Otorhinolaryngol. 2023 Oct;280(10):4433-4444. doi: 10.1007/s00405-023-07961-7. Epub 2023 Apr 12. PMID 37043021
- [Background] Maheo C, Marie A, Torres R, Archutick J, Leclere JC, Marianowski R. Robot-Assisted and Manual Cochlear Implantation: An Intra-Individual Study of Speech Recognition. J Clin Med. 2023 Oct 17;12(20):6580. doi: 10.3390/jcm12206580. PMID 37892718
- [Background] Caversaccio M, Gavaghan K, Wimmer W, Williamson T, Anso J, Mantokoudis G, Gerber N, Rathgeb C, Feldmann A, Wagner F, Scheidegger O, Kompis M, Weisstanner C, Zoka-Assadi M, Roesler K, Anschuetz L, Huth M, Weber S. Robotic cochlear implantation: surgical procedure and first clinical experience. Acta Otolaryngol. 2017 Apr;137(4):447-454. doi: 10.1080/00016489.2017.1278573. Epub 2017 Feb 1. PMID 28145157